CLINICAL TRIAL: NCT04173897
Title: Living Better With Advanced Breast Cancer (LIBERATE) Phase II: Evaluating the Feasibility of a Supportive, Self-management Website in Women Living With Secondary Breast Cancer.
Brief Title: Living Better With Advanced Breast Cancer: Feasibility Evaluation of an Online Supportive Intervention.
Acronym: LIBERATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Breast Cancer Now (Other)
Responsible Party: Principal Investigator, Galina Velikova, Professor Psychosocial Medical Oncology, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NOV2016PhD818
Record Dates: First submitted 2019-10-30; First posted 2019-11-22 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel group, two-arm randomised model using a waiting list control design.
  [A separate single arm study (non-randomised, pre-post design) will run in parallel, recruiting via online channels.]
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): 12 weeks access to LIBERATE online supportive intervention (dose not specified) including symptom monitoring questionnaire component, with questionnaire results integrated within electronic medical records for clinician review.
  Interventions: Other: LIBERATE website
- Waiting list control arm (No Intervention): Care and support as usual; no access to intervention. Placed on waiting list to receive intervention following study completion.

INTERVENTIONS:
Other: LIBERATE website — The LIBERATE intervention is a self-management, symptom monitoring and signposting website tailored to the supportive needs of women living with secondary breast cancer. Components include; holistic health information specific to secondary breast cancer, symptom monitoring and self-management advice, case studies, signposting to services & support and support for family & loved ones.
  Arms: Intervention arm

SUMMARY:
The LIBERATE intervention is a multi-component self-management, symptom monitoring and signposting website tailored to the supportive needs of women living with secondary breast cancer. Overall, this intervention aims to improve quality of life among this growing group of patients through targeted, tailored and accessible information and support.

This randomised waiting list control trial aims to evaluate the feasibility of the clinically integrated LIBERATE intervention. Results of participants' online symptom monitoring questionnaires are integrated with their electronic patient record, enabling clinician review and follow up alongside participants' own self-management activities.

DETAILED DESCRIPTION:
Despite ongoing treatment advances for women living with secondary (metastatic, stage IV, advanced) breast cancer, quality of life (QoL) remains a crucial concern. Patients' diverse psycho-social and supportive needs are widely reported to be poorly understood and inadequately addressed.

The LIBERATE intervention is a multi-component self-management, symptom monitoring and signposting website tailored to the supportive needs of women living with secondary breast cancer.

Phase I of the LIBERATE project informed intervention development though several strands:

1. Semi-structured interviews with patients and health & charity professionals explored the supportive needs and factors affecting the quality of life of women living with secondary breast cancer. This guided the components and content of the online intervention.
2. A systematic review of online interventions in the context of advanced cancer was also conducted. This guided the design and delivery of the online intervention.

The final intervention comprises five components delivered via an interactive website;

* A wide range of holistic health information specific to secondary breast cancer.
* Online symptom monitoring questionnaire generating tailored self-management advice with results available for clinician review.
* Case studies of a diverse range of women living with secondary breast cancer.
* Signposting to services and resources specific to secondary breast cancer.
* Support for others affected by a diagnosis of secondary breast cancer. The overall aims of the LIBERATE intervention are to better address the supportive needs and to improve the quality of life of women living with secondary breast cancer.

Aims and objectives: In this feasibility randomised controlled trial, the investigators plan to test the complete LIBERATE intervention, including the clinical integration of users' symptom monitoring questionnaire results with their electronic medical records.

The investigators aim to examine the feasibility, acceptability and adherence to the online intervention from the perspective of women living with secondary breast cancer and to explore the effect of the intervention on their quality of life and self-efficacy in managing their cancer. The investigators aim to determine effect sizes to inform a potential future larger scale randomised controlled trial.

Eligibility and study design:

Adult females with a diagnosis of secondary breast cancer and access to the internet who are receiving their care at St James' University Hospital, Leeds, will be eligible to take part in this study.

This study will be a prospective randomised controlled feasibility trial using a waiting list control design, repeated measures and mixed methods. Participants will be randomised (following a 1:1 randomisation strategy) to either receive the intervention or to be assigned to a waiting list to receive access to the intervention following study completion. Those on the waiting list will receive care and support as usual during the study period. The investigators aim to recruit a maximum of 30 patients to the study.

Participants in the intervention arm will receive training to navigate the LIBERATE website and complete the online symptom monitoring questionnaires from home. They will be free to use the website as much or as little as they choose over the 12 week study period. They will be reminded to complete a symptom monitoring questionnaire at least once per week. Their health professionals will be able to view the results of their symptom monitoring questionnaires and act on the information accordingly. Alerts will also be sent out to the relevant clinician when patients report any severe symptoms.

All participants (within both the intervention and the waiting list control arm) will complete paper-based self-report questionnaires measuring quality of life and self-efficacy at baseline and at 12 weeks.

A separate single-arm sub study will also recruit approximately 15 women with secondary breast cancer (bringing the overall recruitment target to 45) who are being cared for outside of the Leeds Teaching Hospitals Trust. The aim of this study is to explore whether participants outside of Leeds find symptom monitoring and the overall website useful without the function for linking to their medical records. Participants will fill in questionnaires asking about their QoL and confidence in self-managing their cancer before and after the study.

Study measures:

This study will use a range outcome measures to compare the LIBERATE intervention with care as usual (waiting list control):

Patient reported outcome measures: Validated questionnaires will be used to measure quality of life (EQ-5D-5L and FACT-B) and self-efficacy (CBI-B and SEMCD-6).

Clinical process measures: including number of clinician alerts generated, number of Clinical Nurse Specialist contacts in intervention period, calls to hospital and number of visits to hospital during intervention period.

End of study interviews: semi-structured interviews with participants and health professionals will explore acceptance and experiences of using the LIBERATE intervention.

Overall findings will determine the feasibility and value of a self-management, symptom-monitoring and signposting website as a supportive intervention for women living with and being treated for secondary breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adult females (aged 18 and over).
* Diagnosed with secondary (metastatic, stage IV) breast cancer.
* Access to the internet.

Exclusion Criteria:

* Exhibiting signs of overt psychopathology or cognitive dysfunction.
* Current involvement in other clinical trials involving completion of QoL or other patient reported outcome measures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with self-reported outcome data at 12 weeks. | 12 weeks.
  Patients will complete paper based questionnaires relating to quality of life (FACT-B & EQ-5D-5L) and self-efficacy (B-CBI & SEMCD-6).
Proportion of missing data in self-report outcome questionnaires. | 12 weeks.
  Patients will complete paper based questionnaires relating to quality of life (FACT-B & EQ-5D-5L) and self-efficacy (B-CBI & SEMCD-6).
Appropriateness of each of the self-report outcome questionnaires by assessing ceiling and floor effects (EQ-5D-5L). | 12 weeks
  Descriptive statistics of returned EQ-5D-5L questionnaires.
  The standardised EQ-5D-5L measures health outcomes through a descriptive profile and a visual analogue scale (VAS). The descriptive profile encompasses 5 dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). For each dimension, participants choose one of 5 levels that best describes their health on that day (from 'no problem'= 1 to 'unable/extreme'= 5). The numbers chosen for the five dimensions are combined to give a 5 digit score (minimum score = 11111 maximum score = 55555). The VAS provides participant's rating of their health on a scale from 0 ('the worst health you can imagine') to 100 ('the best health you can imagine').
Appropriateness of each of the self-report outcome questionnaires by assessing ceiling and floor effects (FACT-B). | 12 weeks
  Descriptive statistics of returned FACT-B questionnaires.
Appropriateness of each of the self-report outcome questionnaires by assessing ceiling and floor effects (B-CBI). | 12 weeks
  Descriptive statistics of returned B-CBI questionnaires.
  The 12-item questionnaire Cancer Behaviour Inventory - brief version measures patients' self-efficacy for coping with cancer by asking them to rate their confidence to perform certain behaviours on a scale of 1 (not at all confident) to 9 (totally confident). CBI-B is a single score measure (minimum score = 12, maximum score = 108) with higher scores indicative of greater self-efficacy.
Appropriateness of each of the self-report outcome questionnaires by assessing ceiling and floor effects (SEMCD-6). | 12 weeks
  Descriptive statistics of returned SEMCD-6 questionnaires.
  This 6-item SEMCD-6 measures self-efficacy to manage chronic disease, asking patients to rate their confidence in their abilities to perform a range of self-management tasks. Each of the 6 items are rated on a scale from 1 ('not at all confident') to 10 ('totally confident'). Scores for the scale are calculated as a mean of the 6 items (minimum score = 1, maximum score = 10), with higher scores indicating greater self-efficacy.
Acceptability & use of intervention: Number of symptom monitoring reports generated and qualitative interview data. | 12 weeks
  Number of symptom monitoring reports generated and qualitative interview data.

SECONDARY OUTCOMES:
Estimation of effect size for QOL using participant scores for EQ-5D-5L. | 12 weeks
  Calculation of mean and standard deviation of questionnaire scores to allow for estimation of effect size for QOL.
  [EuroQoL Health Related Quality of Life - 5 Dimensions - 5 Levels (EQ-5D-5L). Descriptive profile minimum score 11111 (no problems across all 5 dimensions), maximum score 55555 (extreme problems). Visual analogue scale rating health from 0 ('worst health imaginable') to 100 ('best health imaginable)].
Estimation of effect size for QOL using participant scores for FACT-B. | 12 weeks
  Calculation of mean and standard deviation of questionnaire scores to allow for estimation of effect size for QOL.
  [Functional Assessment of Cancer Therapy-Breast (FACT-B). Total score ranges from 0 to 123, calculated by adding the scores from each of the 5 subscales. Higher scores reflect better quality of life.]
Estimation of effect size for self-efficacy using participant scores for B-CBI. | 12 weeks
  Calculation of mean and standard deviation of questionnaire scores to allow for estimation of effect size for self-efficacy in managing cancer.
  [Cancer Behaviour Inventory - brief version (B-CBI). Items rated on a scale of 1 (not at all confident) to 9 (totally confident). Single score measure (minimum score =12, maximum score =108), with higher scores indicative of greater self-efficacy].
Estimation of effect size for self-efficacy using participant scores for SEMCD-6. | 12 weeks
  Calculation of mean and standard deviation of questionnaire scores to allow for estimation of effect size for self-efficacy in managing cancer.
  [Self-Efficacy for Managing Chronic Disease scale (SEMCD-6). Items are rated on a scale from 1 ('not at all confident') to 10 ('totally confident'). Scores are calculated as a mean of the 6 items (minimum score =1, maximum score =10), higher scores indicating greater self-efficacy].

CONTACTS AND LOCATIONS:
Locations (1):
- St James University Hospital, Leeds, West Yorkshire, United Kingdom